CLINICAL TRIAL: NCT02328807
Title: Focal Prostate Radio-Frequency Ablation for the Treatment of Prostate Cancer
Brief Title: Focal Prostate Radio-Frequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Trod Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17753
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma; prostate; ENCAGE™; focal bipolar radiofrequency ablation; radiofrequency ablation (RFA); radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- Radio-Frequency Ablation (RFA) (Experimental): Focal Prostate Radio-Frequency Ablation (RFA). Focal bipolar RFA followed by clinical follow-up visits at 6 weeks, 3 months and 6 months.
  Interventions: Procedure: Radio-Frequency Ablation (RFA)

INTERVENTIONS:
Procedure: Radio-Frequency Ablation (RFA) — RFA is a minimally invasive procedure. It is an image-guided technique that heats and destroys cancer cells. In RFA, imaging techniques such as ultrasound or magnetic resonance imaging (MRI) are used to help guide a needle electrode into a cancerous tumor. High-frequency electrical currents are then passed through the electrode, destroying the cancer cells.
  Other Names: ENCAGE™

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of focal (targeted) Radio-Frequency Ablation (RFA) in men with low or intermediate-risk, clinically localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years of age or older
* Diagnosis of adenocarcinoma of the prostate, confirmed by H.L. Moffitt Cancer Center review
* No prior treatment for prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or1
* Prostate Cancer Clinical Stage T2a and below
* PSA <10 ng/ml (this will be the prostatic specific antigen (PSA) level prompting the initial prostate biopsy)
* Prostate size <60 cc on transrectal ultrasound
* Pre-enrollment biopsy parameters (as per H.L. Moffitt C.C. review): Minimum of 10 biopsy cores; Gleason score 6 aor 7; Unilateral cancer (only right-sided or left-sided, not bilateral).

Exclusion Criteria:

* Men less than 18 years of age
* Medically unfit for anesthesia
* Histology other than adenocarcinoma
* Biopsy does not meet inclusion criteria
* Men who have received any hormonal manipulation (antiandrogens; Luteinizing Hormone Releasing Hormone (LHRH) agonist; 5-alpha-reductase inhibitors) within the previous 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Pow-Sang, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six participants were enrolled at Moffitt Cancer Center, August 2015 through July 2017.
Groups:
- Experimental: Radio-Frequency Ablation (RFA) Focal Prostate Ra: Focal Prostate Radio-Frequency Ablation (RFA). Focal bipolar RFA followed by clinical follow-up visits at 6 weeks, 3 months and 6 months.
Period: Overall Study
Arm/Group | Experimental: Radio-Frequency Ablation (RFA) Focal Prostate Ra
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Arm/Group | Experimental: Radio-Frequency Ablation (RFA) Focal Prostate Ra
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 54.66 [50 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Negative Biopsy Rate at 6 Months After Focal Bipolar Radio-Frequency Ablation (RFA)
Description: The primary efficacy endpoint is negative biopsy rate at 6 months after focal bipolar RFA. The point estimate and its 95% confidence interval will be calculated using the exact binominal method.
Time Frame: 6 months
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Radio-Frequency Ablation (RFA) Focal Prostate Ra
Number analyzed (Participants) | 6
Participants
  Negative biopsy | 3
  Recurrence at the ablated area | 2
  Positive biopsy in non-treated contralateral side | 1
Statistical Analysis 1: Comparison: Experimental: Radio-Frequency Ablation (RFA) Focal Prostate Ra; This trail is a single cohort study and no statistical hypothesis test for the primary outcome was planned; Test type: Other; Negative biopsy rate at 6 months after R = 0.667, 95% CI 2-sided [0.223 to 0.957] — Two-sided exact confidence interval was calculated using Clopper-Pearson method

2. Secondary Outcome: Number of Participants With Treatment Related Adverse Events
Description: The type of event using NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 will be identified and graded for severity. The relationship of the adverse event to the therapy or procedure will be determined as follows: Unrelated; Unlikely; Possible; Probable; Definite. For reporting purposes, an adverse event is considered unexpected when either the type of event or severity of the event is not listed in the study consent.
Time Frame: Up to 9 months
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Radio-Frequency Ablation (RFA) Focal Prostate Ra
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Completion of Quality of Life (QOL) Assessment Questionnaires at Six Months
Description: The secondary objective is to evaluate the change from baseline in quality-of-life indicators following focal RFA in patients with low-risk localized prostate cancer. The patients will complete the Expanded Prostate Cancer Index Composite (EPIC), American Urological Association (AUA), Rectal Assessment Scale (RAS), and International Index of Erectile Function (IIEF-5) questionnaires at baseline and 6-month visit. EPIC scores overall 1 (dissatisfied) - 5 (extremely satisfied). AUA scores are o (no prostate issues) - 35 (very severe prostate symptoms). SHIM scores 0 (severe sexual dysfunction) - 25 (no sexual dysfunction) and RAS scores 0 (no bowel issues) - 15 (bad bowel habits)
Time Frame: 6 months
Measure: Median (Full Range); unit: score on a scale
Groups:
- Quality of Life Assessments - Prior to RFA: Quality of Life Assessments prior to focal Prostate Radio-Frequency Ablation (RFA).
- Quality of Life Assessments - After RFA: Quality of Life Assessments after focal Prostate Radio-Frequency Ablation (RFA)
Arm/Group | Quality of Life Assessments - Prior to RFA | Quality of Life Assessments - After RFA
Number analyzed (Participants) | 6 | 6
score on a scale
  SHIM score | 20.66 [11 to 24] | 13 [5 to 20]
  AUA score | 4.66 [1 to 9] | 9 [4 to 19]
  RAS score | 2.33 [1 to 4] | 1.16 [0 to 3]
  EPIC score - Overall Satisfaction | 3.8 [3 to 5] | 3.5 [1 to 5]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Experimental: Radio-Frequency Ablation (RFA) Focal Prostate Ra
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Radio-Frequency Ablation (RFA) Focal Prostate Ra (N=6)
Hematuria (Renal and urinary disorders) | 2 (2)
Other - Blood in semen (Reproductive system and breast disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3)
Other - sciatica (Musculoskeletal and connective tissue disorders) | 1 (2)
Other - prostate sensitivity (Reproductive system and breast disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Renal and urinary disorders - Other, nocturia (Renal and urinary disorders) | 1 (1)
Sinuusitis (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Renal and urinary disorders - Other Dysuria (Renal and urinary disorders) | 1 (2)
Renal and urinary disorders - Other, Burning sensation while urinating (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Accrual ended prior to reaching the study goal due to equipment needing repairs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT02328807/Prot_SAP_000.pdf